CLINICAL TRIAL: NCT05695911
Title: Transfemoral Osseointegrated Prosthesis Limb-Load Symmetry Training
Acronym: TOPLOAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-2116; CDMRPOP220013 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-01-05; First posted 2023-01-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Amputation; Transfemoral Amputation; Osseointegration
Keywords: amputation; osseointegration; rehabilitation; biofeedback

STUDY DESIGN:
Intervention Model Description: Participants will be randomized by ratio of 1:2 in the CTL to EXP group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limb Load Biofeedback Training Intervention (Experimental): The limb-load biofeedback training focuses on altering habitual movement patterns to promote proper prosthetic limb loading with an emphasis on between-limb loading symmetry. Participants randomized to the EXP group will receive 12 biofeedback training sessions (1 in-person, 11 telehealth) tapered over 40 weeks.
  Interventions: Behavioral: Limb Load Biofeedback Training Intervention
- Attention Control Intervention (Placebo Comparator): The CTL group intervention will include the same standard of care rehabilitation sessions as the EXP group and receive the same computer tablets for telehealth sessions as the EXP group. The CTL group will also have attention control educational sessions at the same frequency, timing, and duration as the EXP group limb-load biofeedback sessions (12 total sessions) with the first session being an in-person session at the Week 24. There will be no biofeedback training intervention in the CTL group. As such, there will be no behavioral intervention or wearable sensors provided to the CTL group. The 12 sessions of EXP group limb-load biofeedback training sessions will be replaced by education-only session in the CTL group.
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: Limb Load Biofeedback Training Intervention — Loadsol data will be used to inform the EXP telehealth sessions, as the interventionist guides the participant to self-monitor their movement, problem solve movement patterns that promote asymmetrical limb loading, and create weekly action plans for improving limb load symmetry. Weekly goals will be made in the context of functional task progression over the 40-week intervention.
  Arms: Limb Load Biofeedback Training Intervention
Other: Attention Control — The 12 sessions of EXP group limb-load biofeedback training sessions will be replaced by education-only session in the CTL group. The CTL group sessions will include a review of the standard of care home-exercises, a summary of healthcare visits and falls, and interventionist-delivered education on safety topics (e.g., fall prevention, wound care, assistive device use, home safety).
  Arms: Attention Control Intervention

SUMMARY:
This randomized controlled trial (n=25 enrolled, n=15 expected to complete) will 1) determine the feasibility of a 40-week limb-load biofeedback training intervention, 2) determine if there is an intervention signal of efficacy, and 3) identify functional movement priorities for people with transfemoral osseointegrated (OI) prostheses. A limb-load biofeedback training group (EXP (n=10)) will be compared to a standard of care attention-control group without limb-load biofeedback training (CTL (n=5)). Outcomes will be assessed at standard of care pre-habilitation end (Week 5), standard of care rehabilitation end (Week 24), and one year after OI Stage 2 surgery (Week 64).

DETAILED DESCRIPTION:
This will be a randomized controlled trial with a limb-load biofeedback training (EXP) group and an attention control standard-of-care (CTL) group (2:1 allocation ratio). Outcomes will be assessed prior to surgery (Week 5), start of the limb-load biofeedback training (Week 24), and one year after surgery (Week 64). This Phase I clinical trial will be among the first randomized controlled rehabilitation trials for people with transfemoral OI prostheses. There is an immediate need to better understand the physical health benefits and factors that contribute to poor outcomes for this population. A critical step in developing rehabilitation guidelines is to identify optimal methods for people to regain active lifestyles, best use their prostheses, and avoid secondary comorbidities. This novel limb-load biofeedback training program will provide the empirical evidence necessary to inform post-OI rehabilitation regimens designed to optimize outcomes. Importantly, data from this trial will also guide intervention refinement as the investigators move toward a Phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* Transfemoral unilateral amputation due to traumatic, congenital or cancer related causes
* ≥ 18 years old
* History of severe socket-related skin or residual limb problems
* Schedule for OI prosthesis implantation surgery

Exclusion Criteria:

* Vascular amputation etiology
* Substance abuse
* Unstable heart condition
* Acute systemic infection
* Cognitive impairment (Montreal Cognitive Assessment [MoCA] score <24)
* Active cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | Week 64
  Intervention feasibility is measured by retention rate, the percentage of people that complete the study. A score can range between 0 and 100 percent with 100 percent meaning all randomized participants completed the study.
Intervention Participant Acceptability | Week 64
  Acceptability of an intervention is the perception among stakeholders (e.g., patients and clinicians) that the intervention is agreeable or satisfactory. To measure participant acceptability, the investigators will use the Acceptability of Intervention Measure, a 30 four-item survey of stakeholder perception of intervention acceptability that asks participants to provide their approval as well as intervention appeal, likability, and agreeability. The scores range from 1 (completely disagree) to 5 (completely agree). The investigators expect the Acceptability of Intervention Measure score (average of the four items on a 1-5 scale) for the EXP group to be at least 4 (agree).
Intervention Fidelity | Week 64
  This will be evaluated based on whether EXP group interventionists deliver the intervention as planned and quantified in three ways: adherence, delivery quality, and patient engagement. The investigators will use the overall results of these three fidelity components to create a total score. Fidelity scores are reported as a percentage from 0 to 100 with 100 representing full fidelity. The investigators will consider >85% fidelity (average across all three components) to intervention delivery as a positive result.
Change in Cumulative Loading | Week 5, Week 64
  Free-living physical activity will be objectively monitored over a 10-day period using an activPAL micro accelerometer-based sensor (PAL Technologies, Glasgow, UK). Interlimb cumulative loading will be measured as a product of daily step count and ground reaction force impulse. Cumulative loading = (Daily Steps/2)*ground reaction force impulse.
Change in Multi-Domain Biomechanics during Tasks of Increasing Biomechanical Demand | Week 5, Week 64
  Bilateral hip movement patterns (joint angles), muscle forces, and joint reaction forces will be calculated during functional tasks of increasing biomechanical demand (walking, sitting, stepping, turning) using a combination of motion capture and subject-specific musculoskeletal models. Whole-body motion capture will be collected from 70 reflective markers (Fs=120 Hz) (Vicon, Centennial, CO) with ground reaction forces simultaneously collected from six embedded force platforms (Fs=2,160 Hz) (Bertec, Columbus, OH). A subject-specific musculoskeletal model will be created using OpenSim software.

SECONDARY OUTCOMES:
Change in World Health Organization-Disability Assessment Schedule 2.0 | Week 5, Week 24 and Week 64
  Self reported questionnaire measuring disability in adults age 18 years and older. Final scores range from 0 (no disability) to 100 (full disability).
Change in Activities Specific Balance Confidence Scale | Week 5, Week 24 and Week 64
  Self reported measure of balance confidence. Final scores range from 0% (no confidence in balance) to 100% (complete confidence in balance).
Change in Prosthetic Limb Users Survey of Mobility | Week 5, Week 24 and Week 64
  A 12 item self report questionnaire measuring participants mobility when using a prosthesis. Final scores range from 12 to 60 points with higher scores indicating greater mobility.
Change in Patient Specific Function Scale | Week 5, Week 24 and Week 64
  Self reported questionnaire measuring the ability of the participant to do 3 self identified activities. Scores of each of the 3 activities range from 0 (unable to perform) to 10 (able to perform without difficulty). Total scores range from 0 to 30 points, with higher scores indicating higher function.
Change in Self Selected Gait Speed | Week 5 and Week 64
  Test to quantify walking ability as it is associated with health outcomes, fall risk, and mobility levels and is also a frequent indicator of intervention effectiveness. The time it takes each participant to walk 5-meters (after 3-meter acceleration zone, followed by 3-meter deceleration zone). The self selected gait speed will be averaged over three trials.
Change in 30 Second Sit - Stand Test | Week 5, Week 64
  Test to assess lower-extremity strength and endurance. The number of times the participant can rise from sitting in 30 seconds.
Change in Colorado Osseointegrated Limb Donning and Timed Up and Go Test | Week 5, Week 64
  A specific test to measure physical function and balance. The time it takes a participant to don their prosthesis, rise from sitting, walk 10 feet and turn, walk back to the chair and return to seated position.

CONTACTS AND LOCATIONS:
Overall Officials: Cory Christiansen, PT PHD, Principal Investigator — University of Colorado, Denver
Locations (1):
- CU Physical Therapy, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will publish the trial results data on the ClinicalTrials.gov website, on which the clinical trial will be registered. Sharing of data will include the potential of sharing raw data generated from all clinical assessments under a data-sharing agreement.
Supporting Information: ICF
Time Frame: The investigators will publish the trial results within one year of testing the final participant.
Access Criteria: User registration will be required to access/download any data and will require agreement to conditions of use in accordance with CDMRP Policy on Sharing Data and Research Resources.